CLINICAL TRIAL: NCT01330290
Title: A Multi-site, Non-interventional, Cross-sectional Evaluation of the Caregivers' and the Physicians' Preferred Route of Administration and the Physicians' Rationale for the Choice of Neupro® in Patients With Parkinson Requiring Caregiver Support
Brief Title: Caregivers' and Physicians' Treatment Preference in Parkinson Patients Treated With Neupro® Requiring Caregiver Support
Acronym: CARE-ACT
Status: Completed | Type: Observational
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: SP0939
Record Dates: First submitted 2011-03-18; First posted 2011-04-06 (Estimated); Results first posted 2013-12-10 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-11

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Rotigotine; Neupro®; Parkinson; Treatment preference; Care-giving
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Neupro® Treatment: Routine treatment (2, 4, 6, 8, 10, 12, 14, 16 mg/24 hours) as per approved label in European Union (EU)/in accordance with the terms of the local marketing authorization for Neupro®
  Interventions: Drug: Neupro®

INTERVENTIONS:
Drug: Neupro® — Neupro patches were prescribed by the treating physician according to the Summary of the Product Characteristics. Patients with idiopathic Parkinson's Disease (iPD) were treated for at least 1 month with a combination of Levodopa (L-DOPA) or other oral iPD medication and Neupro by the time the questionnaire was completed.
  Other Names: Rotigotine

SUMMARY:
The study objective is to evaluate advantages and disadvantages of Neupro® versus oral anti-Parkinson medication by caregivers and physicians in idiopathic Parkinson's Disease patients requiring caregiver support in nursing home or outpatient care settings.

ELIGIBILITY:
Inclusion Criteria:

* Only patients having signed the consent form regarding study information, data transfer and data use
* The patients suffer from idiopathic Parkinson's Disease (iPD) treated with a combination of L-dopa or another oral iPD drug and Neupro® for at least one month
* The patients require caregiver support documented as per medical records (e.g. based on German level of care intensity 1 or greater)
* The decision to prescribe Neupro® must have been made by the physician independent of his/her decision to include the patient in the study

Exclusion Criteria:

* Patients not fulfilling the inclusion criteria
* And according to Summary of Product Characteristics (SmPC): Hypersensitivity to the active substance or to any of the excipients, magnetic resonance tomography (MRT) or cardioversion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Idiopathic Parkinson's Disease (iPD) patients treated with a combination of L-dopa or other oral iPD drug and Neupro® for at least one month and requiring caregiver support documented as per medical records
  Every consecutive, eligible patient to be treated with Neupro® as per physician's decision
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2011-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (54):
- Germany (54):
  - 52, Abensberg
  - 53, Alzenau in Unterfranken
  - 18, Beelitz-Heilstätten
  - 42, Bensheim
  - 24, Berlin
  - 27, Berlin
  - 37, Celle
  - 58, Cologne
  - 17, Dillingen
  - 48, Dresden
  - 32, Eisenach
  - 39, Erbach im Odenwald
  - 43, Erfurt
  - 60, Essen
  - 5, Gelnhausen
  - 40, Gelsenkirchen
  - 31, Göttingen
  - 38, Guelders
  - 29, Hagen
  - 57, Halle
  - 6, Halle
  - 28, Hamm
  - 47, Hanover
  - 7, Herborn
  - 55, Hoppegarten
  - 59, Jena
  - 50, Karlstadt am Main
  - 44, Königsbrück
  - 51, Lappersdorf
  - 8, Lohr
  - 4, Marktheidenfeld
  - 45, Merzig
  - 36, Minden
  - 34, Mittweida
  - 35, Mühldorf
  - 25, München
  - 41, München
  - 30, Münster
  - 49, Neuburg am Inn
  - 21, Neumarkt
  - 13, Niederschöna
  - 9, Oschatz
  - 54, Schorndorf
  - 2, Schriesheim
  - 1, Stralsund
  - 12, Stratroda
  - 15, Stuttgard
  - 33, Stuttgart
  - 20, Ulm
  - 14, Unterhaching
  - 22, Weil am Rhein
  - 11, Westerstede
  - 23, Wolfach
  - 56, Wolfratshausen

REFERENCES:
- [Derived] Sieb JP, Themann P, Warnecke T, Lauterbach T, Berkels R, Grieger F, Lorenzl S. Caregivers' and physicians' attitudes to rotigotine transdermal patch versus oral Parkinson's disease medication: an observational study. Curr Med Res Opin. 2015 May;31(5):967-74. doi: 10.1185/03007995.2015.1030376. PMID 25772231
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients participating in this study were in need of care either by family members at home or by professional nurses in outpatient care or nursing homes. The Participant Flow refers to the Enrolled Set (ES). All patients who were entered into the database are included in the Enrolled Set (ES).
Pre-assignment Details: The physicians were instructed to select idiopathic Parkinson's Disease (iPD) patients with documented need of care with caregivers/nurses who attended patients at home as caregiving family members or as professional nurses in outpatient care or nursing homes.
Groups:
- Neupro® Treatment: Routine treatment (2, 4, 6, 8, 10, 12, 14, 16 mg/24 hours) as per approved label in European Union (EU)/in accordance with the terms of the local marketing authorization for Neupro®
  Neupro® : Neupro patches were prescribed by the treating physician according to the Summary of the Product Characteristics. Patients with idiopathic Parkinson's Disease (iPD) were treated for at least 1 month with a combination of Levodopa (L-DOPA) or other oral iPD medication and Neupro by the time the questionnaire was completed.
Period: Overall Study
Arm/Group | Neupro® Treatment
Started | 148
Completed | 148 (As this is a cross-sectional study, the terms completed/not completed are not applicable.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Characteristics refer to the Enrolled Set (ES). All patients who were entered into the database are included in the Enrolled Set (ES).
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 148
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 131
Age Continuous [Mean (Standard Deviation); unit: years] | 74.61 (8.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 88
Region of Enrollment [Number; unit: participants]
  Germany | 148
Weight [Mean (Standard Deviation); unit: kilogram] | 73.43 (14.71)
Height [Mean (Standard Deviation); unit: centimeters] | 168.39 (10.28)
Type of care-giving: Patient lives at nursing home [Number; unit: participants]
  No | 108
  Yes | 16
  Missing | 24

OUTCOME MEASURES:

1. Primary Outcome: Mean Score of the Caregivers' Rating of Neupro® Compared to Oral Anti-Parkinson Medication
Description: The caregivers were asked to fill out a questionnaire composed of 7 questions covering caregiving aspects. The mean score is calculated from the scores for the single responses which are rated from 'great disadvantages' to 'great advantages' and scored on a 5-point scale from -2 to +2.
  Each caregiver could have assessed one or multiple participants. The scores from each caregiver were averaged over all participants they assessed, and the final mean score was calculated from the averaged assessments of the caregivers.
Time Frame: Questionnaire completed at a single time-point during the run of the cross-sectional study (16 months). Suitable patients suffer from idiopathic iPD treated with a combination of l-dopa or another oral iPD drug and Neupro® for at least one month.
Population: The Analysis Population refers to the Full Analysis Set (FAS). The Full Analysis Set (FAS) comprises all patients with at least 1 assessment in the physicians' or caregivers'/nurses' questionnaires. The average assessment of all patients assessed by a distinct caregiver was calculated and used for analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Averaged Assessments
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 147
Number analyzed (Averaged Assessments) | 126
units on a scale | 1.32 (0.67)

2. Primary Outcome: Mean Score of the Physicians' Rating of Neupro® Compared to Oral Anti-Parkinson Medication
Description: The physicians were asked to fill out a questionnaire composed of 10 questions covering medical and caregiving aspects. The mean score is calculated from the scores for the single responses which are rated from 'great disadvantages' to 'great advantages' and scored on a 5-point scale from -2 to +2.
  Each physician could have assessed one or multiple participants. The scores from each physician were averaged over all participants they assessed, and the final mean score was calculated from the averaged assessments of the physicians.
Time Frame: as for outcome 1
Population: The Analysis Population refers to the Full Analysis Set (FAS). The Full Analysis Set (FAS) comprises all patients with at least 1 assessment in the physicians' or caregivers'/nurses' questionnaires. The average assessment of all patients assessed by a distinct physician was calculated and used for analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Averaged Assessments
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 147
Number analyzed (Averaged Assessments) | 40
units on a scale | 1.46 (0.32)

3. Secondary Outcome: Assessment of the Physicians' Rationale for the Choice of Neupro® Due to Substance in Idiopathic Parkinsons Disease Patients Requiring Caregiver Support
Description: The physician was asked if he / she prescribed Neupro® due to substance in idiopathic Parkinson's Disease patients requiring caregiver support. The possible answers were "applicable" and "not applicable".
Time Frame: as for outcome 1
Population: The Analysis Population refers to the Full Analysis Set (FAS). The Full Analysis Set (FAS) comprises all patients with at least 1 assessment in the physicians' or caregivers'/nurses' questionnaires.
Measure: Number; unit: participants
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 147
participants
  Applicable | 89
  Not applicable | 57
  Missing | 1

4. Secondary Outcome: Assessment of the Physicians' Rationale for the Choice of Neupro® Due to Application Form in Idiopathic Parkinsons Disease Patients Requiring Caregiver Support
Description: The physician was asked if he / she prescribed Neupro® due to application form in idiopathic Parkinson's Disease patients requiring caregiver support. The possible answers were "applicable" and "not applicable".
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 147
participants
  Applicable | 139
  Not applicable | 7
  Missing | 1

5. Secondary Outcome: Score for the Physicians' Rating of Neupro® Compared to Oral Anti-Parkinson Medication in Relation to Dysphagia in Patients With Dysphagia
Description: This individual question from the caregivers' questionnaire was to be assessed from "major disadvantages" to "major advantages", and the corresponding answer was to be evaluated according to a 5-point rating scale using a score from -2 to +2.
  Each physician could have assessed one or multiple participants. The scores from each physician were averaged over all participants they assessed, and the final mean score was calculated from the averaged assessments of the physicians.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Averaged Assessments
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 147
Number analyzed (Averaged Assessments) | 30
units on a scale | 1.59 (0.82)

6. Secondary Outcome: Score for the Physicians' Rating of Neupro® Compared to Oral Anti-Parkinson Medication in Relation to Nausea and/or Vomiting in Patients With Nausea and/or Vomiting.
Description: This individual question from the physicians' questionnaire was to be assessed from "major disadvantages" to "major advantages", and the corresponding answer was to be evaluated according to a 5-point rating scale using a score from -2 to +2.
  Each physician could have assessed one or multiple participants. The scores from each physician were averaged over all participants they assessed, and the final mean score was calculated from the averaged assessments of the physicians.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Averaged Assessments
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 147
Number analyzed (Averaged Assessments) | 30
units on a scale | 1.48 (0.54)

7. Secondary Outcome: Score for the Physicians' Rating of Neupro® Compared to Oral Anti-Parkinson Medication in Relation to Control of Compliance
Description: as for outcome 6
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Averaged Assessments
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 147
Number analyzed (Averaged Assessments) | 40
units on a scale | 1.36 (0.59)

8. Secondary Outcome: Score for the Physicians' Rating of Neupro® Compared to Oral Anti-Parkinson Medication in Relation to Multiple Medication in Patients With Multiple Medication
Description: as for outcome 6
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Averaged Assessments
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 147
Number analyzed (Averaged Assessments) | 40
units on a scale | 1.48 (0.60)

9. Secondary Outcome: Score for the Physicians' Rating of Neupro® Compared to Oral Anti-Parkinson Medication in Relation to Surgery Requiring General Anaesthesia
Description: as for outcome 6
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Averaged Assessments
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 147
Number analyzed (Averaged Assessments) | 35
units on a scale | 1.87 (0.32)

10. Secondary Outcome: Score for the Physicians' Rating of Neupro® Compared to Oral Anti-Parkinson Medication in Relation to Dose Adaption
Description: as for outcome 6
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Averaged Assessments
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 147
Number analyzed (Averaged Assessments) | 27
units on a scale | 1.35 (0.75)

11. Secondary Outcome: Score for the Physicians' Rating of Neupro® Compared to Oral Anti-Parkinson Medication With Regard to Independency of Food Administration
Description: as for outcome 6
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Averaged Assessments
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 147
Number analyzed (Averaged Assessments) | 40
units on a scale | 1.50 (0.44)

12. Secondary Outcome: Score for the Physicians' Rating of Neupro® Compared to Oral Anti-Parkinson Medication With Regard to Sleeping Patients
Description: as for outcome 6
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Averaged Assessments
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 147
Number analyzed (Averaged Assessments) | 40
units on a scale | 1.37 (0.58)

13. Secondary Outcome: Score for the Physicians' Rating of Neupro® Compared to Oral Anti-Parkinson Medication in Relation to Risk of Interaction With Other Treatments
Description: as for outcome 6
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Averaged Assessments
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 147
Number analyzed (Averaged Assessments) | 40
units on a scale | 1.15 (0.63)

14. Secondary Outcome: Score for the Physicians' Rating of Neupro® Compared to Oral Anti-Parkinson Medication in Relation to Resorption
Description: as for outcome 6
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Averaged Assessments
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 147
Number analyzed (Averaged Assessments) | 40
units on a scale | 1.64 (0.55)

15. Secondary Outcome: Score for the Caregivers' Rating of Neupro® Compared to Oral Anti-Parkinson Medication in Relation to Dysphagia in Patients With Dysphagia
Description: This individual question from the caregivers' questionnaire was to be assessed from "major disadvantages" to "major advantages", and the corresponding answer was to be evaluated according to a 5-point rating scale using a score from -2 to +2.
  Each caregiver could have assessed one or multiple participants. The scores from each caregiver were averaged over all participants they assessed, and the final mean score was calculated from the averaged assessments of the caregivers.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Averaged Assessments
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 147
Number analyzed (Averaged Assessments) | 68
units on a scale | 1.44 (0.94)

16. Secondary Outcome: Score for the Caregivers' Rating of Neupro® Compared to Oral Anti-Parkinson Medication in Relation to Nausea and/or Vomiting in Patients With Nausea and/or Vomiting
Description: as for outcome 15
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Averaged Assessments
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 147
Number analyzed (Averaged Assessments) | 60
units on a scale | 1.50 (0.91)

17. Secondary Outcome: Score for the Caregivers' Rating of Neupro® Compared to Oral Anti-Parkinson Medication in Relation to Control of Compliance
Description: as for outcome 15
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Averaged Assessments
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 147
Number analyzed (Averaged Assessments) | 127
units on a scale | 1.33 (0.93)

18. Secondary Outcome: Score for the Caregivers' Rating of Neupro® Compared to Oral Anti-Parkinson Medication in Relation to Multiple Medication in Patients With Multiple Medication
Description: as for outcome 15
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Averaged Assessments
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 147
Number analyzed (Averaged Assessments) | 123
units on a scale | 1.49 (0.79)

19. Secondary Outcome: Score for the Caregivers' Rating of Neupro® Compared to Oral Anti-Parkinson Medication With Regard to Independency of Food Administration
Description: as for outcome 15
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Averaged Assessments
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 147
Number analyzed (Averaged Assessments) | 126
units on a scale | 1.54 (0.77)

20. Secondary Outcome: Score for the Caregivers' Rating of Neupro® Compared to Oral Anti-Parkinson Medication With Regard to Sleeping Patients
Description: as for outcome 15
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Averaged Assessments
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 147
Number analyzed (Averaged Assessments) | 124
units on a scale | 1.19 (0.91)

21. Secondary Outcome: Score for the Caregivers' Rating of Neupro® Compared to Oral Anti-Parkinson Medication in Relation to Care-giving Efforts
Description: as for outcome 15
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Averaged Assessments
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 147
Number analyzed (Averaged Assessments) | 126
units on a scale | 1.03 (0.98)

ADVERSE EVENTS:
Time Frame: All Adverse Drug Reactions (ADRs) were collected at the time of data collection.
Description: The physicians were asked to list on the corresponding registration form all Adverse Events (AEs) that were documented at the time of data collection and were asked to assess if the causal relationship to the application of Neupro was classified as Yes (=ADR) or No.
Arm/Group | Neupro® Treatment
Serious Adverse Events (participants affected / at risk) | 0/148
Other Adverse Events (participants affected / at risk) | 1/148
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neupro® Treatment (N=148)
Palpitations (Cardiac disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days